CLINICAL TRIAL: NCT00938288
Title: A Phase I Study to Determine the Pharmacokinetic Profile, Safety and Tolerability of a Single Dose (50IU/kg) of KW-3357 in Subjects With Congenital Antithrombin Deficiency.
Brief Title: A Study of KW-3357 in Congenital Antithrombin Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3357-EU-001; EudraCT number 2008-005504-16
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Congenital Antithrombin Deficiency
Keywords: Antithrombin; Thrombosis; Pharmacokinetics; Hereditary Antithrombin Deficiency; Congenital Antithrombin Deficiency
MeSH Terms: conditions — Thrombosis; Antithrombin III Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Single group
  Interventions: Drug: KW-3357

INTERVENTIONS:
Drug: KW-3357 — 50IU/mL, IV single dose

SUMMARY:
The aim of this study is to determine the pharmacokinetics, safety and tolerability of KW-3357 in asymptomatic subjects with congenital antithrombin deficiency.

DETAILED DESCRIPTION:
Patients with Congenital Antithrombin Deficiency are at increased risk of venous thrombosis and pulmonary embolism especially when undergoing certain high risk procedures. Antithrombin replacement therapy is often administered during these periods, with or without low molecular weight heparin. Prior to assessing the efficacy of KW-3357, a new recombinant human antithrombin, the present study will determine it's pharmacokinetics, safety and tolerability in subjects who have Congenital Antithrombin Deficiency but who are currently asymptomatic and not undergoing a high-risk procedure. Up to 16 evaluable subjects will be enrolled at multiple investigational sites over a period of approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years of age with congenital Antithrombin deficiency (AT activity ≤60% of normal) in a stable condition without evidence of acute thromboembolic events
* Signed IEC-approved Informed Consent Form
* Subjects must not have received an infusion of Antithrombin for at least 14 days before Screening
* Patients of reproductive potential must agree to follow accepted birth control methods during the study

Exclusion Criteria:

* Subjects who are classified as morbidly obese (defined by the presence of a body mass index >40 kg/m2)
* Subjects who have participated in a study with an investigational drug within 30 days of Screening or within 5.5 times the elimination half-life of the investigational drug before Screening, whichever period is greater
* Subjects with any clinically relevant medical history or current condition or physical findings, ECG, or laboratory values which could interfere with the objectives of the study or the safety of the subject
* Subjects using non-steroidal anti-inflammatories, fondaparinux sodium, dabigatran or rivaroxaban or who are expected to be treated with these drugs during the study
* Subjects who have concomitant nephrotic syndrome
* Female subjects who are pregnant or lactating
* Subjects who are taking heparin, low molecular weight heparin and/or oral anticoagulants, with the exception of vitamin K antagonists (eg, warfarin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12-22 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic profile of a single dose (50 IU/kg) of KW 3357 in subjects with congenital AT deficiency | July 2011

SECONDARY OUTCOMES:
To determine the safety and tolerability of a single dose (50 IU/kg) of KW-3357 in subjects with congenital AT deficiency | July 2011

CONTACTS AND LOCATIONS:
Overall Officials: Beverley Hunt, FRCP, FRCPath MD, Principal Investigator — St Thomas' Hospital, London, UK
Locations (8):
- Department of Haemotogy, Haemastasy, Oncology and Stem Cell Transplantation, Hannover Medical School, Hanover, Germany
- Sweden (2):
  - Center for Thrombosis and Haemostasis, Malmo University Hospital, Malmo
  - Dept Obst Gyn/Section for Women and Child Health/Clinical Trial Unit, Karolinska University Hospital, Stockholm
- United Kingdom (5):
  - Treliske, Haematology Clinic, Royal Cornwall Hospital, Truro, Cornwall
  - Bristol Haemophia Care Centre, Bristol Haemotology and Oncology Centre, Bristol
  - Department of Haemotology, Glasgow Royal Infirmary, Glasgow
  - Kings College, Dept of Haematology, Lupus & Pathology Guy's and St Thomas Trust, St Thomas Hospital, Ctr for Haemostasis and Thrombosis (the Haemophia Reference Ctr), London
  - University College London Hospital NHS Trust, London